CLINICAL TRIAL: NCT05826496
Title: Characterization of Immunological Parameters in Blood from Healthy Participants Before and After High- to Moderate-intensity Aerobic Exercise
Brief Title: Exercise-induced Effects on Immune Parameters in Healthy Participants
Acronym: INHALE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Per thor Straten (Other)
Responsible Party: Sponsor-Investigator, Per thor Straten, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-23006672; IN2301 (Other: CCIT)
Record Dates: First submitted 2023-03-23; First posted 2023-04-24 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Acute exercise; Virus-specific T cells; High-intensity interval training; T cell; Acute stress response; NK cell; Inflammation; Exercise immunology; Catecholamines
MeSH Terms: conditions — Inflammation | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: HLA-A2 positive participants complete one acute bout of supervised aerobic high-intensity exercise
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise (Experimental): HLA-A2 positive participants will perform one bout of high-intensity interval training.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The supervised high-intensity interval training is conducted on bicycle ergometers at 85-95% maximal workload. The high-intensity interval sequences will be separated by two steady state sequences. Blood samples are collected at baseline, 2 min and 60 min post-exercise.

SUMMARY:
Exercise has been shown to influence the immune system and, for example, improve anti-viral immune response. However, knowledge of how exercise impacts the immune system is still lacking. Therefore, the goal of this clinical study is to perform a comprehensive multi-parameter analysis of immunological parameters in healthy participants before and after one bout of high-intensity aerobic exercise. The primary endpoint of this study is to determine the exercise-induced changes of anti-viral T cell immunity in peripheral blood against common and recurrent viruses.

Up to 70 healthy participants in the age between 18 and 75 will be recruited. The first visit will be for prescreening the health status, answering questionnaires and providing a capillary blood sample for HLA screening. HLA-A2 positive participants will continue on the trial with a VO2 max test for Visit 2 and the supervised aerobic medium- to high-intensity (90% VO2 max) exercise session for Visit 3. Peripheral blood samples will be taken pre-exercise, within 2 minutes post-exercise and 60 minutes post-exercise.

These findings may pave the way to define serum markers or cellular immunological traits that provide new insight into how exercise promotes powerful and sustained cellular immune responses.

DETAILED DESCRIPTION:
Numerous physiological parameters are influenced by exercise, including marked changes on numerous markers of the immune system. It has been shown that exercise lowers systemic low-grade inflammation, and there are indications that exercise improves the ability to combat infections and vaccination-induced immune responses.

Exercise has been repeatedly shown to mobilize immune cells into peripheral blood - most pronouncedly prototype killer cells of both the innate and adaptive immune system namely Natural Killer (NK) and T cells. Both cell types are critical in immune responses against viral infections and are also key effector cells in anti-cancer immune responses. Even more so, previously activated NK and T cells are selectively mobilized, potentially providing the background for exercise-mediated stronger anti-viral immunity.

In this study, the blood samples will be used to study global viral T cell reactivity against chronic [Cytomegalovirus (CMV) and Ebstein-Barr virus (EBV)] and recurrent [Influenza (flu) and SARS-CoV-2] viruses and detect their exact frequencies in peripheral blood. Since the technique is optimized for HLA*A2:01 positive individuals, this study will include a prescreening to match this tissue type. Adding more complexity to the acquired data, further analyses include but are not limited to phenotyping by CyTOF and flow cytometry as well as Luminex immune assays.

The current study will provide important insight into how the immune system is influenced by acute medium-to high-intensity exercise. These findings may have important implications for vaccine development, prevention in frail and at-risk populations, cancer prevention and cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have the ability to speak and read English and/or Danish.
* Agree to avoid alcohol, nonprescription drugs, and strenuous exercise for 24 hours prior VO2 max test and exercise intervention.
* Signed informed consent.

Exclusion Criteria:

* Autoimmune disease requiring active treatment.
* A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications. Inhaled or topical steroids and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted
* Use of medication known to affect the immune system (regular use of ibuprofen/aspirin or beta-blockers).
* Any systemic infections with fever within the last 4 weeks before the exercise intervention.
* Use of any illegal drugs (e.g., cocaine, amphetamine).
* Conditions with high risk for complications during exercise: Unstable medical disease, condition, or history of serious or concurrent illness; any medical condition that might be aggravated by exercise training or that cannot be controlled, including, but not restricted to congestive heart failure (NYHA class III-IV), unstable angina pectoris, implantable cardioverter defibrillator (ICD), or myocardial infarction within 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Virus-specific T cell responses | 6 months
  Investigate the number of virus-reactive CD8+ T cells at baseline, within 2 minutes after cessation and 60 minutes after cessation of the exercise bout in peripheral blood using DNA-barcoded peptide-MHC multimer assay.

SECONDARY OUTCOMES:
Phenotypes of exercise-mobilized immune cells | 6 months
  The investigators will assess the phenotype of immune cells in peripheral blood at baseline, within 2 minutes after cessation and 60 minutes after cessation of the exercise bout using Flow Cytometry and CyTOF.
Circulating soluble markers | 1 year
  The investigators will analyse a panel of serum markers that reflect the effect of high-intensity exercise and its timely dynamics using Luminex and ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Holmen Olofsson, PhD, Principal Investigator — CCIT, Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No